CLINICAL TRIAL: NCT00258739
Title: A Phase II, Randomized Study With Docetaxel-gemcitabine Followed by Radiotherapy vs Concomitant Treatment (Radiotherapy and Carboplatine-docetaxel) Followed by Docetaxel-gemcitabine Versus Docetaxel-gemcitabine Followed by Concomitant Treatment (Radiotherapy and Carboplatine-docetaxel) in Stage III NSCLC
Brief Title: Docetaxel in Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAX_ES1_209
Record Dates: First submitted 2005-11-23; First posted 2005-11-28 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel; Carboplatin; Radiotherapy; Gemcitabine

ARMS (2):
- 1 (Experimental): Concomitant radiotherapy and carboplatin-docetaxel followed by docetaxel-gemcitabine
  Interventions: Drug: Docetaxel + carboplatin + radiotherapy + docetaxel + gemcitabine
- 2 (Experimental): docetaxel-gemcitabine followed by concomitant radiotherapy with carboplatin-docetaxel
  Interventions: Other: Docetaxel + gemcitabine + carboplatin + radiotherapy

INTERVENTIONS:
Drug: Docetaxel + carboplatin + radiotherapy + docetaxel + gemcitabine — Docetaxel 20 mg/m²/week with carboplatin AUC 2/week and concomitant radiotherapy up to 60 Gy. Further on, 2 Docetaxel cycles and gemcitabine according to arm 2.
  Arms: 1
Other: Docetaxel + gemcitabine + carboplatin + radiotherapy — Docetaxel 40 mg/ m² days 1, 8, 21 and 28 with gemcitabine 1200 mg/ m² days 1, 8, 21 and 28 followed by concomitant treatment with docetaxel 20 mg/m²/week with carboplatin AUC 2/week and concomitant radiotherapy up to 60 Gy (2 Gy/day, 5 days per week and for 6 weeks).
  Arms: 2

SUMMARY:
Primary objective:

* To classify the 2 study groups, according to the tumoral response.

Secondary objectives:

* To evaluate the percentage of focused control per year.
* To calculate the time until progression.
* To evaluate the safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Non small cell lung cancer confirmed by histology or by cytology.
* IIIB stage, except if existing pleural discharge, upper cava vein syndrome or supraclavicular affectation
* General stage 0-1 at the ECOG scale
* Loss of weight less than 5% in the 3 previous months from diagnose.
* Pulmonary function and gasometry results: FEV1 > 30% or 1 l, DLCO (diffusing capacity of the lung for carbon monoxide) > 30%, PCO2 < 45 mmHg and PO2 > 60 mmHg.
* Normal medullar function (hemoglobin > 11 g/dl, total WBC > 1,5 x 10^9/l, platelets > 100 x 10^9/l)
* Appropriate renal and hepatic functions
* CTScan
* Anticonceptive method
* Available laboratory test (maximum 1 month before)

Exclusion criteria:

* Pleural discharge, upper cava vein syndrome or supraclavicular affectation.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2001-10; Primary Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Response rate in each arm measured according to RECIST criteria | Throughout the whole study

SECONDARY OUTCOMES:
Percentage of local-regional control within a year | Throughout the first year
Time to progression defined as the period of time elapsed between the randomization date and the progression or death date | Throughout the whole study
Toxicity measured by CALGB criteria and RTOG/EORTC criteria | Throughout the whole study
Global surveillance measured as the period of time elapsed between randomization and death date. | Throughout the whole study duration

CONTACTS AND LOCATIONS:
Overall Officials: José Mª Taboada, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Barcelona, Spain